CLINICAL TRIAL: NCT05371899
Title: Absorption, Metabolism and Excretion of [14C]Chiauranib in Patients With Small Cell Lung Cancer
Brief Title: Mass Balance Study of [14C]Chiauranib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR109
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Chiauranib; pharmacokinetic characteristics; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiauranib (Other): Take 50 mg ChiauranibCioroni capsules orally on an empty stomach once a day, every day; except on the eighth day 8, when you start taking Cioroni capsules liquid, take a single oral dose of ~50 mg/about 100 Ci of [14C]Chiauranib suspensionCioroni solution once on an empty stomach.
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — Take Chiauranib 50mg orally once daily

SUMMARY:
Chiauranib , which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

DETAILED DESCRIPTION:
Chiauranib , which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

This trial is a material balance study of [14C]Chiauranib in participants with small cell lung cancer, with the goal of learning more about the drug's absorption, metabolism, and excretion in the human body, as well as monitoring the subjects' safety after treatment. Chiauranib's scientific foundation for future progress.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18 Years to 75 Years
* Cytologically or histologically confirmed small cell lung cancer
* After normal therapy, disease progression or returnrecurrence
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 3 months
* Laboratory criteria are as follows:

  * Complete blood count: absolute neutrophil count (ANC) ≥1.5×10^9/L ; platelets ≥75×10^9/L; hemoglobin (Hb) ≥80g/L ;
  * Biochemistry test: total bilirubin≤1.5×ULN; alanine aminotransferase (ALT) , aspartate aminotransferase(AST)≤2.5×ULN(ALT,AST≦5×ULN if liver involved); serum creatinine(cr)≤1.5×ULN;
  * Coagulation test: International Normalized Ratio (INR) < 1.5.
* All patients must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Patients experiencing neurological symptoms due to liver or brain metastases
* Patients with hemoptysis or tumor invading around important blood vessels and hemoptysis during the screening period
* Pleural fluid, ascites, pericardial effusion with clinical symptoms and need to be drained during the screening period
* Patients with second primary cancer, except: adequately treated basal cell or squamous cell skin cancer, curatively treated in-situ cancer of the cervix, unless received curative treatment and with documented evidence of no recurrence during the past five years
* Sunitinib, bevacizumab, anlotinib, apatinib, endostat, and other Aurora kinase inhibitors or VEGF/VEGFR inhibitors were used to treat this small cell lung cancer
* Patients have used any anti-cancer therapy, including, chemotherapy, immunotherapy, target therapy, and other anti-tumor treatments within 14 days before the first dose, Patients have used adiotherapy within 14 days before the first dose
* Patients received major surgical operations within 28 days before the first dose, or patients with serious non-healing wounds, ulcer or fracture at the time of screening
* With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy
* Abnormal and clinically significant ophthalmic examination
* Patients with uncontrolled or significant cardiovascular disease, including:

  * Grade II or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (NYHA Classification) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage.
  * Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al).
  * History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male),QTc≥470ms（female）at screening.
  * patient's treatment record of using at least 2 antihypertensive drugs at the same Within 14 days before the first dose, or uncontrolled hypertension (> 140/90 mmHg) during the screening period.
* Lung disease that seriously affects ventilation or diffusing function during the screening period
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction, After small bowel resection,etc), or undergone gastrectomy, or history of gastrointestinal perforation
* Unhealed diarrhea prior to dosing, or 4 or more episodes of diarrhea within 7 days prior to planned dosing, or habitual diarrhea
* Habitual constipation persists after treatment
* During the screening period, when the urine protein in the routine urine test is ≥2+, a 24-hour urine protein quantitative test should be carried out. Protein ≥2+, quantitative examination <1g/24h can be enrolled
* Active bleeding within 2 months before the first dose, or anticoagulant drugs are being taken during the screening period, or the investigator judges that there is a high risk of bleeding during the screening period
* History of deep vein thrombosis or pulmonary embolism within 6 months before the first dose
* Active infections that require systemic treatment (oral, intravenous infusion) during the screening period
* With clinically significant UTI or genital infection, or with a history of complicated UTI
* Positive for any one of hepatitis B surface antigen, hepatitis B e antigen, hepatitis C antibody, HIV antibody, syphilis antibody and new crown screening
* Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study
* Allergic to cioroni capsules and its excipients
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism(CYP3A, CYP1A2 and CYP2D6)within 30 days prior to drug administration of the study medication
* Any other condition which is inappropriate for the study according to investigators' judgment
* Binge drinking or drinking greater than 14 units of alcohol per week in the 6 months prior to screening; or alcohol breath test results ≥ 20 mg/dl during the screening period
* Smoking more than 5 cigarettes per day or habitual use of nicotine-containing products within 2 months before screening, or unable to quit during the trial
* Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages and inability to withdraw during the trial
* Drug abuse or drug abuse that affects the evaluation of test results, or a positive urine drug test during the screening period
* Women of childbearing potential not willing to use and utilize an adequate method of contraception (such as intrauterine device, contraceptive and condom) throughout treatment and for at least 12 weeks after the last dose; pregnant or breastfeeding women; the result of urine pregnancy test was positive at screening; Man participants not willing to use and utilize an adequate method of contraception throughout treatment
* Engaged in work requiring prolonged exposure to radioactive conditions; or participated in radiopharmaceutical labeling experiments
* Difficulty of venous blood collection
* Volunteer in any other study within 3 months prior to drug administration, or Volunteer in 3 times or more studies
* Blood donation or lost more than 400mL blood within 3 months prior to the study, or Received blood transfusions within 1 month
* Other situations that the researchers considered unsuitable to enroll the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Tmax | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Time to maximum concentration
Cmax | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Maximum concentration
AUC | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Area under the plasma concentration-time curve
t1/2 | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Half life
MRT | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Mean resident time
Whole blood/plasma concentration (B/P) ratios for total radioactivity | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Whole blood/plasma concentration (B/P) ratios for total radioactivity
Cumulative amount of radioactivity recovered in urine, feces, and in total | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Cumulative amount of radioactivity recovered in urine, feces, and in total
Percent of Metabolite in plasma, urine and feces | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Percent of Metabolite in plasma, urine and feces

SECONDARY OUTCOMES:
percentage of AEs | The sample collection for the last subject was done, and the safety inspection was performed，assessed up to 22 days
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Huang, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No